CLINICAL TRIAL: NCT03638648
Title: Multi Gene Detection Tool Based Recurrence Score-guiding Chemotherapy in Non-pathologic Complete Response HR Positive and HER2 Negative Breast Cancer After Neoadjuvant Treatment
Brief Title: Recurrence Score-guiding Chemotherapy in Non-pCR HR Positive HER2 Negative Breast Cancer After Neoadjuvant Therapy
Acronym: RSBNAT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RS-NAT01
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
Keywords: breast cancer; neoadjuvant; multiple gene detection
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low risk Capecitabine (Active Comparator): Patients after neoadjuvant chemotherapy evaluated as non-pCR have multiple gene test based low recurrence risk receiving capecitabine.
  Interventions: Drug: Capecitabine
- Low risk control (No Intervention): Patients after neoadjuvant chemotherapy evaluated as non-pCR have multiple gene test based low recurrence risk NOT receiving any additional chemotherapy.
- High risk Capecitabine (Experimental): Patients after neoadjuvant chemotherapy evaluated as non-pCR have multiple gene test based high recurrence risk receiving capecitabine.
  Interventions: Drug: Capecitabine
- High risk control (No Intervention): Patients after neoadjuvant chemotherapy evaluated as non-pCR have multiple gene test based high recurrence risk NOT receiving any additional chemotherapy.

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 2500mg/m2/day, d1-d14, every 3 weeks a cycle for 8 cycles
  Other Names: additional chemotherapy
  Arms: High risk Capecitabine; Low risk Capecitabine

SUMMARY:
The luminal subtype of breast cancer means hormone receptor positive, human epidermal growth factor receptor 2 negative (HR+HER2-), which counted 60%-70% of breast cancer but achieve low pathologic complete response (pCR) rate (7.5%-15%) in neoadjuvant chemotherapy. It is controversial whether additional chemotherapy after surgery is necessary for those non-pCR HR+HER2- patients. Multiple gene is a mature diagnose tool for recurrence score in adjuvant treatment strategy. This study is to investigating the value of multi gene detection tool based recurrence score for guiding additional chemotherapy after surgery in HR+HER2- non-pCR breast cancer.

DETAILED DESCRIPTION:
This study is designed as stratified cluster randomized, parallel-control research. The HR+HER2- breast cancer patients after neoadjuvant chemotherapy (including anthracyclines and taxane, at least 6 cycles) assessed non-pCR are recruited, receiving multiple gene test before neoadjuvant treatment and after surgery. After enrollment, the patients were stratified according to multiple gene test based recurrence risk level (High risk or Low risk) and then randomized into two groups respectively in each cluster: receiving additional chemotherapy (Capecitabine) group or negative control group. The primary endpoint is 2-year disease free survival. The second endpoint is 5-year disease free survival (DFS), 2-year overall survival (OS), 5-year OS, safety of additional chemotherapy. The exploratory endpoint is the variety of multiple gene test based recurrence risk after neoadjuvant chemotherapy in non-pCR patients.

ELIGIBILITY:
Inclusion Criteria:

1. Invasive breast cancer at the first diagnosed
2. Clinical stage cT1-4cN0-3M0 (AJCC 8th), receiving neoadjuvant chemotherapy at least 6 cycles
3. Neoadjuvant chemotherapy regimen should include anthracyclines and taxane
4. Primary tumor HR+(ER+ or PR+) and HER2 negative before neoadjuvant chemotherapy
5. Pathological evaluation non-pCR after neoadjuvant chemotherapy (residual invasive cancer in primary tumor)

Exclusion Criteria:

1. Metastasis, recurrent breast cancer or receiving other treatment before neoadjuvant chemotherapy
2. Pregnant breast cancer
3. IHC or FISH test of primary tumor confirmed HER2 positive at anytime
4. Complete fewer than 6 cycles chemotherapy before surgery
5. Deficiency of surgery after neoadjuvant
6. Contraindication of chemotherapy or surgery

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
2-year DFS | 2 years after randomized
  disease-free survival rate in 2 years

SECONDARY OUTCOMES:
5-year DFS | 5 years after randomized
  disease-free survival rate in 5 years
2-year OS | 2 years after randomized
  overall survival rate in 2 years
5-year OS | 5 years after randomized
  overall survival rate in 5 years
Aside effect | 5 years
  any aside effect induced by additional chemotherapy (Capecitabine)

OTHER OUTCOMES:
variety of multiple gene based recurrence score | half year after randomized
  recurrence score before and after neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Xingfei Yu, MD, Principal Investigator — Zhejiang Cancer Hospital

IPD SHARING:
Plan to Share IPD: No